CLINICAL TRIAL: NCT00562627
Title: Efficacy of Multimodal Peri- and Intraarticular Drug Injections in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Ulrich Johannes Spreng, Asker and Baerum Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-003030-41; EudraCT 2007-003030-41; REK 1.2007.1603
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Results first posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee arthroplasty; local infiltration analgesia; TKA; epidural analgesia; operation; surgery
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Ropivacaine; Epinephrine; Ketorolac; Ketorolac Tromethamine; Morphine; Fentanyl; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LIA IV (Experimental): Local infiltration analgesia with ropivacaine and adrenaline and intravenous ketorolac and morphine
  Interventions: Drug: ropivacaine; Drug: adrenaline; Drug: ketorolac; Drug: morphine
- LIA IA (Experimental): Local infiltration analgesia with ropivacaine, adrenaline and ketorolac and morphine
  Interventions: Drug: ropivacaine; Drug: adrenaline; Drug: ketorolac; Drug: morphine
- EDA (Active Comparator): standard continuous epidural analgesia
  Interventions: Drug: adrenaline; Drug: fentanyl; Drug: bupivacaine

INTERVENTIONS:
Drug: ropivacaine — intraoperative and 1. postoperative day
  Other Names: Naropin
  Arms: LIA IA; LIA IV
Drug: adrenaline — intraoperative LIA (IV and IA) and continuous EDA
  Other Names: Adrenalin; (epinephrine)
Drug: ketorolac — intraoperative and 1. postoperative day
  Other Names: Toradol
  Arms: LIA IA; LIA IV
Drug: morphine — intraoperative
  Other Names: Morfin
  Arms: LIA IA; LIA IV
Drug: fentanyl — continuous postoperatively
  Arms: EDA
Drug: bupivacaine — continuous postoperatively
  Other Names: Marcain
  Arms: EDA

SUMMARY:
Total knee arthroplasty (TKA) is associated with moderate to severe postoperative pain, causing patient discomfort, mobilisation and hospital discharge.

The aim of this study is to:

1. Compare analgetic efficacy of to types of local infiltration analgesia in total knee arthroplasty.
2. Compare analgetic efficacy of local infiltration analgesia with continuous epidural analgesia.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is increasingly common in the treatment of knee osteoarthritis. TKA is associated with moderate to severe postoperative pain, causing patient discomfort, mobilisation and hospital discharge.

Continuous epidural analgesia is often used for controlling pain after TKA. Recent studies describe a new method for pain control after total knee arthroplasty which consists of local infiltration with local anesthetics and adrenaline. This infiltrations can be combined with ketorolac and/or morphine. The aim of this study is to:

1. Compare analgetic efficacy of to types of local infiltration analgesia in total knee arthroplasty.
2. Compare analgetic efficacy of local infiltration analgesia with continuous epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* patients at least 18 years of age
* scheduled for elective total knee arthroplasty
* ASA I-III
* signed written informed consent

Exclusion Criteria:

* age < 18
* ASA > III
* moderate or severe cardiac disease, bronchial asthma
* allergy against ropivacaine, ketorolac or morphine
* analgetic abuse
* pregnancy or nursing women
* severe psychiatric disease
* moderate to severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich J Spreng, MD, Principal Investigator — Asker and Baerum Hospital
Locations (1):
- Asker and Baerum Hospital, Rud, Norway

REFERENCES:
- [Derived] Spreng UJ, Dahl V, Hjall A, Fagerland MW, Raeder J. High-volume local infiltration analgesia combined with intravenous or local ketorolac+morphine compared with epidural analgesia after total knee arthroplasty. Br J Anaesth. 2010 Nov;105(5):675-82. doi: 10.1093/bja/aeq232. Epub 2010 Aug 24. PMID 20736233

RESULTS

PARTICIPANT FLOW:
Groups:
- LIA IV (Local Infiltration Analgesia, Intravenous): Local infiltration analgesia with 150 mg ropivacaine and 0.5 mg adrenaline and intravenous 30 mg ketorolac and 5mg morphine
- LIA IA, (Local Infiltration Analgesia, Intra-articular): Local infiltration analgesia with 150 mg ropivacaine, 0.5 mg adrenaline and 30 mg ketorolac and 5 mg morphine
- Epidural: continuous epidural analgesia with fentanyl 2 ug/ml, bupivacaine 1mg/ml and epinephrine 1 ug/ml
Period: Overall Study
Arm/Group | LIA IV (Local Infiltration Analgesia, Intravenous) | LIA IA, (Local Infiltration Analgesia, Intra-articular) | Epidural
Started | 34 | 34 | 34
Completed | 33 | 33 | 33
Not Completed | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LIA IV (Local Infiltration Analgesia, Intravenous) | LIA IA, (Local Infiltration Analgesia, Intra-articular) | Epidural | Total
Number analyzed (Participants) | 34 | 34 | 34 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 17 | 47
  >=65 years | 18 | 20 | 17 | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 66.5 (11) | 67.2 (8.9) | 65.8 (10.7) | 66.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 23 | 65
  Male | 13 | 13 | 11 | 37
Region of Enrollment [Number; unit: participants]
  Norway | 34 | 34 | 34 | 102

OUTCOME MEASURES:

1. Secondary Outcome: Opioid Use
Description: Morphine used by patient controlled analgesia. Amount of used morphine during the first 48 hours after surgery were documented in the CRF by the pain nurses.
Time Frame: 48 hours postoperative
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | LIA IV (Local Infiltration Analgesia, Intravenous) | LIA IA, (Local Infiltration Analgesia, Intra-articular) | Epidural
Number analyzed (Participants) | 33 | 33 | 33
mg | 77 (39) | 49 (36) | 54 (43)
Statistical Analysis 1: Comparison: LIA IV (Local Infiltration Analgesia, Intravenous) vs LIA IA, (Local Infiltration Analgesia, Intra-articular) vs Epidural; Test type: Superiority or Other; p = 0.009, ANOVA

2. Primary Outcome: Pain at Rest (VAS)
Description: VAS (pain at rest) 0-100 mm. VAS 0 mm means no pain and VAS 100 mm means maximal pain.
Time Frame: 48 hours postoperative
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | LIA IV (Local Infiltration Analgesia, Intravenous) | LIA IA, (Local Infiltration Analgesia, Intra-articular) | Epidural
Number analyzed (Participants) | 33 | 33 | 33
Units on a scale | 18 (15) | 12 (13) | 30 (29)
Statistical Analysis 1: Comparison: LIA IV (Local Infiltration Analgesia, Intravenous) vs LIA IA, (Local Infiltration Analgesia, Intra-articular) vs Epidural; Test type: Superiority or Other; p = 0.001, ANOVA

3. Secondary Outcome: Time to Readiness for Discharge
Description: Each postoperative day, discharge readiness was assessed by an orthopaedic surgeon, a pain nurse, a ward nurse, and a physiotherapist according to the following criteria: no evidence for surgical complications, VAS pain at rest ≤30 mm which is controlled by oral analgesics, ability to eat and drink, ability to walk with elbow crutches, and ability to climb ≥8 stairs.
Time Frame: up to 10 days postoperative
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LIA IV (Local Infiltration Analgesia, Intravenous) | LIA IA, (Local Infiltration Analgesia, Intra-articular) | Epidural
Number analyzed (Participants) | 33 | 33 | 33
days | 4 (1.3) | 3.5 (0.7) | 5.5 (1.6)
Statistical Analysis 1: Comparison: LIA IV (Local Infiltration Analgesia, Intravenous) vs LIA IA, (Local Infiltration Analgesia, Intra-articular) vs Epidural; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Arm/Group | LIA IV (Local Infiltration Analgesia, Intravenous) | LIA IA, (Local Infiltration Analgesia, Intra-articular) | Epidural
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 1/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LIA IV (Local Infiltration Analgesia, Intravenous) (N=33) | LIA IA, (Local Infiltration Analgesia, Intra-articular) (N=33) | Epidural (N=33)
Knee infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes